CLINICAL TRIAL: NCT04985162
Title: Comparison of the Effects of Ordinary and Differential Learning Based Physiotherapy on Subjects With Ischemic Stroke Torso Control, Balance and Gait in the Second Phase of Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Laura Smilgiene, Laura Smilgiene, physiotherapist, Lithuanian University of Health Science, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2021-07-26; First posted 2021-08-02 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were divided into intervention group and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group (n=10) received differential learning based physiotherapy program: 3 times a week ordinary physiotherapy, 2 times a week differential learning based on physiotherapy, total 3 weeks
  Interventions: Other: Intervention group
- Control (Active Comparator): Control group (n=10) received ordinary physiotherapy program 5 times a week, total 3 weeks
  Interventions: Other: Control group

INTERVENTIONS:
Other: Intervention group — Differential learning based physiotherapy to improve torso control, balance and gait
  Arms: Intervention
Other: Control group — Ordinary physiotherapy program
  Arms: Control

SUMMARY:
The purpose of this study was to assess the effect or ordinary and differential learning based physiotherapy for torso control, balance and gait on subjects with ischemic stroke in the second phase of rehabilitation

DETAILED DESCRIPTION:
Ischemic stroke is still the second most common cause of death and one of the leading causes of disability worldwide. Half of all individuals with ischemic stroke do not regain lost body functions until the end of life. Individuals with ischemic stroke are most likely to have impaired cognitive, sensory, and motor functions, but the greatest challenge for health care professionals is impaired motor skills caused by motor nerve cell damage. In order to minimize the degree of disability, it is important to respond quickly to a person's condition. Because it has been shown that lost functions can be taken over by adjacent, non-stroke-affected areas of the cerebral cortex, early rehabilitation is a key factor that can help prevent function limitation by acting in conjunction with spontaneous recovery of body function.

The aim of the study is to assess the effect or ordinary and differential learning based physiotherapy for torso control, balance and gait on subjects with ischemic stroke in the second phase of rehabilitation.

The study was approved by Committee on Biomedical Research Ethics of Kaunas Region (2020-06-30 No.BEC-KN(B)-263).

ELIGIBILITY:
Inclusion Criteria:

* Patients rehabilitated in Neurorabilitation Departmen of Lithuanian University of Health sciences hospital Kauno Kliniko in the second stage of rehabilitation;
* Stroke for the first time;
* 45-74 m. age;
* Able to go with aids;
* Voluntary consent to participate in the study.

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Torso control assessment scale | Baseline to 3 weeks
  The torso control rating scale evaluates torso functions in a variety of locations, whether standing, sitting or performing a mobility assessment task. Each task was scored from 0 to 3 points: 0 - cannot perform task, 3 - can perfom task independently. Total test score is 36 and a higher total score meant a better trunk function.
Berg balance test | Baseline to 3 weeks
  The Berg scale is used to assess a subject's static and dynamic balance. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4. The maximum obtainable score is 56. 0 points -are awarded to answers portraying the lowest level of function while 4 points are awarded to the highest level of function.
Dynamic gait index is used to assess the likelihood of falling. A four-point ordinal scale, ranging from 0-3 points. Total maximum score is 24 points. 0 points indicates the lowest level of function and 3 points - the highest level of function. | Baseline to 3 weeks
  Dynamic gait index assessed the gait model, provided information about the person's balance while walking

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences, Department of Rehabilitation, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided